CLINICAL TRIAL: NCT07187076
Title: Body Awareness in Geriatric Individuals
Brief Title: Body Awareness Therapy in Geriatric Individuals: Role of Biopsychosocial Dynamics
Acronym: Body Awareness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Seda Karaca, phd, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025/429
Record Dates: First submitted 2025-09-15; First posted 2025-09-22 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Geriatric
Keywords: body awareness; geriatric

STUDY DESIGN:
Intervention Model Description: This study follows a parallel-group randomized controlled interventional model, designed to assess the impact of a Body Awareness-Based Exercise Program (BAEP) on both physical function and psychological well-being in older adults. It adopts a single-blind approach in which the outcome assessor remains unaware of group allocations to reduce detection bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- body awareness (Experimental): body awareness exercises
  Interventions: Behavioral: body awareness

INTERVENTIONS:
Behavioral: body awareness — Body Awareness Therapy (BAT) is a somatic-based, movement-centered therapeutic approach that aims to improve individuals' physical, emotional, and psychological well-being by enhancing conscious awareness of bodily sensations, posture, breathing, movement, and internal states.
  Originating from Scandinavian physiotherapy models - particularly the work of Berit Heir Bunkan, Roxendal, and Dropsy - BAT integrates principles from:
  Proprioceptive neuromuscular retraining
  Mindfulness-based movement
  Sensorimotor integration
  Psychomotor physiotherapy
  BAT is not simply a set of physical exercises, but a neuropsychophysical method designed to promote:
  Postural control and alignment
  Somatic grounding and bodily coherence
  Emotional regulation through movement
  Enhanced interoception (awareness of internal bodily states)

SUMMARY:
Population aging is one of the most significant global health trends of the 21st century. As life expectancy increases, so do the physical and psychological challenges faced by older adults. Aging is associated with a progressive decline in muscle mass and strength (sarcopenia), reduced mobility, impaired balance, altered gait mechanics, and an increased risk of falls. In addition to these physical changes, older individuals frequently experience psychosocial issues such as anxiety, depression, social isolation, and diminished quality of life.

Conventional physiotherapy programs for elderly individuals typically focus on balance, strength, and mobility training. While these are undeniably effective, they may not fully address the mind-body connection, proprioceptive awareness, and emotional regulation, which are equally important for maintaining overall well-being and functional independence. Recently, body-awareness-based exercise methods have gained attention for their potential to bridge this gap by fostering conscious movement, breath awareness, and improved self-regulation.

Body Awareness Therapy (BAT), also referred to in the literature as "body awareness-based physiotherapy," is a therapeutic approach that combines gentle physical movements, breathing exercises, postural control, and relaxation techniques. It has been used effectively in various populations, including individuals with chronic pain, mental health disorders, neurological conditions, and musculoskeletal impairments. However, limited evidence exists on its potential applications in geriatric populations, particularly concerning its influence on both physical functioning and psychological well-being.

This study was designed to investigate the effects of a structured Body Awareness-Based Exercise Program (BAEP) on older adults, focusing on its potential to improve physical function (balance, gait, mobility, strength) and psychological outcomes (anxiety, depression, and life satisfaction).

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the effects of an 8-week body awareness-based exercise intervention on:

Physical function: including balance, lower extremity strength, and functional mobility.

Psychological well-being: including anxiety, depression, and perceived life satisfaction.

The secondary objective was to assess the feasibility and adherence to the intervention in an elderly population.

3. Methodology 3.1 Study Design

This was a prospective, single-blinded, randomized controlled trial involving two parallel groups:

Experimental Group: received standard physiotherapy plus Body Awareness-Based Exercise Program (BAEP)

Control Group: received only standard physiotherapy care.

The total duration of the intervention was 8 weeks.

3.2 Participants

Participants were recruited from a university-affiliated geriatrics outpatient clinic. A total of 32 elderly individuals, aged 60-80 years, who met the inclusion criteria were randomly allocated to either group using a computerized randomization tool.

Inclusion Criteria

Aged 60-80 years

Able to ambulate independently or with minimal assistance

MMSE score ≥ 24 (cognitively competent)

Medically cleared for physical activity

No history of falls in the last 6 months

Willingness to participate and sign informed consent

Exclusion Criteria

Severe visual, vestibular, or neurological impairments

Uncontrolled cardiovascular or pulmonary conditions

Cognitive impairment (MMSE < 24)

Acute illness or musculoskeletal injury

Ongoing participation in another structured exercise program

Missing more than 2 consecutive sessions

3.3 Sample Size

A priori power analysis (using G*Power 3.1) indicated that a minimum sample of 16 participants per group (total N = 32) would be required to detect a clinically significant change in the 6-Minute Walk Distance (6MWD), with 80% power and an alpha of 0.05.

4. Interventions 4.1 Standard Physiotherapy Program

Both groups participated in a baseline physiotherapy program consisting of:

Respiratory Exercises:

Diaphragmatic breathing

Thoracic expansion (segmental breathing)

Aerobic Training:

Treadmill or overground walking, progressive intensity

Strengthening Exercises:

Resistance band-based lower limb exercises

Balance and Gait Training

Energy conservation techniques and ADL regulation

This was implemented 6 days per week for 8 weeks. Three sessions were supervised, and the remaining were home-based, with telephone monitoring for adherence.

4.2 Body Awareness-Based Exercise Program (BAEP)

Participants in the experimental group additionally received a 1-hour BAEP session once per week, conducted by a physiotherapist with 4 years of experience in the method. The protocol was based on principles by Roxendal and Dropsy, incorporating:

Movement-Based Awareness Training (MBAT)

Breath-focused floor and standing exercises

Pelvic mobility and spinal rotation

Postural alignment and midline recognition

Relaxation and proprioceptive feedback enhancement

All exercises were initiated in supine position to minimize energy demand and maximize sensory feedback. The program was progressively adapted to each individual's comfort and capacity.

Participants were encouraged to keep a body awareness diary to reflect on sensations, posture, and psychological states post-session.

5. Outcome Measures 5.1 Baseline and Post-Intervention Assessments

All assessments were conducted at week 0 and repeated at week 8.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years and older, living independently in the community.

Capable of walking independently or with minimal assistance.

Exclusion Criteria:

* Diagnosed with severe cognitive impairment (MMSE < 24) or dementia.

Having unstable cardiovascular, pulmonary, or neurological conditions in the past 6 months.

Inability or unwillingness to participate in scheduled sessions or comply with the study protocol.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 73 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-14 (Actual)

PRIMARY OUTCOMES:
Body Awareness Questionnaire (BAQ) | 8 weeks
  valuates the participant's level of body awareness and interoceptive attention, which is the core target of your intervention.
Change in Functional Exercise Capacity | Baseline and 8 weeks after the start of the intervention
  The primary outcome will be the change in the distance walked during the 6-Minute Walk Test (6MWT), which is a validated and widely used measure of functional exercise capacity in older adults. Participants will be asked to walk at their own pace in a standardized indoor corridor for 6 minutes, and the total distance (in meters) will be recorded. The test will be conducted following the American Thoracic Society guidelines.

CONTACTS AND LOCATIONS:
Locations (1):
- Guneysu Physiotherapy School, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
due to patients' rights